CLINICAL TRIAL: NCT07291401
Title: Neoadjuvant Chemoradiotherapy Combined Cith Iparomlimab and Tuvonralimab (QL1706) Therapy for Locally Advanced Rectal Cancer：a Single-center, Prospective, Randomized, Phase II Clinical Trial
Brief Title: Radiotherapy Plus CAPOX, and Iparomlimab and Tuvonralimab (QL1706) as Neoadjuvant Therapy for LARC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025056
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer Patients
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A patients received radiotherapy, chemotherapy, and immunotherapy. During the first week of radiotherapy, they received one cycle of CAPOX concurrent chemoradiotherapy. Two weeks after the completion of radiotherapy, they continued with four cycles of CAPOX combined with QL1706 immunotherapy.
  Interventions: Combination Product: lparomlimab and Tuvonralimab Injection and CPAOX and radiotherapy
- Group B (Experimental): Group B patients received radiotherapy and chemotherapy. After completing the concurrent radiotherapy and chemotherapy, they rested for 2-3 weeks before completing 3 cycles of CAPOX consolidation chemotherapy.
  Interventions: Combination Product: CPAOX and radiotherapy

INTERVENTIONS:
Combination Product: lparomlimab and Tuvonralimab Injection and CPAOX and radiotherapy — Neoadjuvant chemoradiotherapy + immunotherapy: Pelvic radiotherapy (IMRT), 36 Gy/12 fractions/3 weeks; adaptive radiotherapy booster of 5-6 Gy/2 fractions is permitted for residual lesions. During the first week of radiotherapy, one cycle of CAPOX regimen concurrent chemoradiotherapy is administered (oxaliplatin, 100 mg/m2, D1, IV drip; capecitabine, 850 mg/m2, BID, oral on the day of radiotherapy). Two weeks after radiotherapy, four cycles of IT-CAPOX regimen immunotherapy combined with chemotherapy are continued (epaloliposide (QL1706) 5 mg/kg, D1, IV drip; oxaliplatin, 130 mg/m2, D1, IV drip; capecitabine, 1000 mg/m2, BID, PO, D1-14, Q3W). Two to three weeks after the completion of immunotherapy and chemotherapy, a comprehensive follow-up evaluation of efficacy is conducted, and surgical treatment is planned.
  Arms: Group A
Combination Product: CPAOX and radiotherapy — Neoadjuvant concurrent chemoradiotherapy: Pelvic radiotherapy, IMRT 45-50.4 Gy/25-28 F, for a total of 5-6 weeks. During radiotherapy, administer oral capecitabine concurrent chemoradiotherapy (capecitabine, 850 mg/m2, BID, orally on the day of radiotherapy). After radiotherapy, rest for 2-3 weeks, then complete 3 cycles of CAPOX consolidation chemotherapy (oxaliplatin, 130 mg/m2, D1, IV drip; capecitabine, 1000 mg/m2, BID, PO, D1-14, Q3W). 2-3 weeks after the completion of consolidation chemotherapy, conduct a comprehensive follow-up assessment of the efficacy, and surgical treatment is planned.
  Arms: Group B

SUMMARY:
This study is a single-center, prospective, randomized, double-arm, Phase II clinical trial designed to evaluate the efficacy of radiotherapy combined with CAPOX, and Iparomlimab and Tuvonralimab (QL1706) as neoadjuvant therapy for locally advanced rectal cancer. Additionally, the study seeks to explore the relationship between biomarkers in blood and tumor tissue and treatment efficacy.

Eligible participants (locally advanced rectal cancer) were randomly assigned in a 1:1 ratio to two groups.

Participants will:

Group A patients received radiotherapy, chemotherapy, and immunotherapy. During the first week of radiotherapy, they received one cycle of CAPOX concurrent chemoradiotherapy. Two weeks after the completion of radiotherapy, they continued with four cycles of CAPOX combined with QL1706 immunotherapy.

Group B patients received radiotherapy and chemotherapy. After completing the concurrent radiotherapy and chemotherapy, they rested for 2-3 weeks before completing 3 cycles of CAPOX consolidation chemotherapy.

Two to three weeks after the completion of neoadjuvant therapy in groups A and B, the efficacy was evaluated, and a decision was made on whether to proceed with surgery or watchful waiting based on the efficacy.

DETAILED DESCRIPTION:
Improving the tumor downstaging rate and complete response rate of neoadjuvant therapy remains a key focus and hot topic in clinical research. Neoadjuvant immunotherapy has been recommended by clinical guidelines for locally advanced rectal cancer (LARC) with DNA mismatch repair deficiency/high microsatellite instability (dMMR/MSI-H), achieving a pCR rate as high as 60-70%. However, the efficacy of immunotherapy in locally advanced rectal cancer with microsatellite stable disease (pMMR/MSS), which accounts for the vast majority, remains controversial. Recent phase II studies have shown that combining chemotherapy and immunotherapy with long-course or short-course radiotherapy may further improve the pCR rate to 30-40% compared to traditional concurrent chemoradiotherapy. In a study by Professor Zhang Zhen's team at Fudan University, short-course radiotherapy combined with consolidation or induction chemotherapy and immunotherapy even achieved a cCR rate exceeding 50%. A meta-analysis published in 2025 also showed that in pMM locally advanced rectal cancer patients receiving neoadjuvant radiotherapy combined with immunotherapy, patients receiving short-course radiotherapy combined with PD-1 inhibitors or concurrent immunoradiotherapy showed better treatment outcomes, while the toxic side effects were tolerable. However, these studies have small sample sizes, lack consistency in drug use and study design, and have insufficient levels of evidence, requiring further exploration and verification.

This study will explore the efficacy and safety of neoadjuvant chemoradiotherapy combined with erato combination antibody for the treatment of locally advanced pMMR rectal cancer through a prospective phase II randomized controlled clinical trial, aiming to provide a reference for achieving higher cCR/pCR rates and preservation of anal function in patients with locally advanced rectal cancer.

Specifically, the study will assess the pathological complete response (pCR) rate two weeks after neoadjuvant therapy, the clinical complete response (cCR) rate under the "watch-and-wait" strategy, R0 resection rate, tumor regression grade (TRG), and sphincter preservation rate. Additionally, the study will evaluate the 3-year disease-free survival (DFS) and overall survival (OS) following dual-inhibitor combined neoadjuvant chemoradiotherapy. The safety and tolerability of this combination therapy will also be comprehensively assessed based on NCI-CTCAE 4.03 criteria.

ELIGIBILITY:
Inclusion Criteria:

* (1) The patient is histologically diagnosed with rectal adenocarcinoma. (2) Age ≥18 years, <75 years (3) Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 (4) AJCC stage of rectal cancer: cT3-4N0M0 or TanyN1-2M0 (5) The lower margin of the rectal tumor is ≤10cm from the anus. (6) At least one evaluable lesion based on RECIST 1.1 assessment. (7) Subjects should have adequate bone marrow and liver and kidney function reserves:

  * Neutrophils ≥1.5×10⁹/L, platelets ≥75×10⁹/L, and hemoglobin ≥9 g/dL

    * Total bilirubin ≤1.5×Upper limit of normal (UNL); ASAT (SGOT) and/or ALAT (SGPT) ≤2.5×UNL (≤5×UNL if liver metastasis occurs); alkaline phosphatase ≤2.5×UNL (≤5×UNL if liver metastasis occurs, ≤10×UNL if bone metastasis occurs); LDH <1500 U/L

      * Creatinine clearance (calculated according to the Cockcroft and Gault formula) >60 mL/min or serum creatinine ≤1.5×UNL; (8) Voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

* (1) Histopathological examination confirms the presence of other pathological types, such as squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma, etc.

  (2) Pathological examination confirms microsatellite highly unstable dMMR/msi-H (3) Presence of intestinal obstruction, intestinal perforation, bleeding, or other conditions requiring emergency surgery (4) History of pelvic radiotherapy (5) Comorbid malignant tumors (excluding cervical carcinoma in situ that has been cured for more than 2 years) (6) Receiving any other anti-tumor treatment (chemotherapy, radiotherapy, surgery, targeted therapy, immunotherapy) or participating in other new drug clinical trials within the past 4 weeks (7) Presence of the following cardiovascular and cerebrovascular diseases or risks:
  1. Myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (Class 2 or above as determined by the New York Heart Association functional classification) within 6 months prior to randomization, symptomatic or poorly controlled arrhythmia
  2. 3 years prior to first use of the drug a. History of pulmonary embolism or other serious thromboembolism within the past month
  3. Presence of aortic aneurysm, aortic dissection aneurysm, internal carotid artery stenosis or other major vascular diseases that may endanger life or require surgery within the past 6 months
  4. History of myocarditis or cardiomyopathy or current examination suggests myocarditis
  5. Left ventricular ejection fraction (LVEF) <50%
  6. Complete left bundle branch block, third-degree atrioventricular block (8) Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment, or an autoimmune disease that the investigator judges may relapse or is planned for treatment. The following are excluded:

  <!-- -->

  1. Skin diseases that do not require systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema)
  2. Hypothyroidism caused by autoimmune thyroiditis that requires only stable doses of hormone replacement therapy
  3. Type I diabetes that requires only stable doses of insulin replacement therapy
  4. Childhood asthma that has completely resolved and requires no intervention in adulthood
  5. The investigator determines that the disease will not recur without external triggering factors (9) Known or suspected active pulmonary tuberculosis (10) Subjects with active hepatitis B, inactive or asymptomatic hepatitis B virus (HBV) carriers (HBsAg positive) with HBV DNA > 500 IU/mL or > 2500 copies/mL), and subjects with active hepatitis C should be excluded. Inactive or asymptomatic carriers of hepatitis B who are treated and stable and meet the criteria of HBV DNA ≤500 IU/mL or ≤2500 copies/mL are eligible for enrollment. Subjects with cured hepatitis C who are HCVAb positive and HCV RNA negative are eligible for enrollment. (11) Subjects who require systemic treatment with glucocorticoids (>10 mg/day prednisone or equivalent dose) or other immunosuppressive drugs within 14 days prior to randomization. The following are exceptions:

  a. Inhaled, ophthalmic, or topical corticosteroids are permitted if there is no active autoimmune disease.

  b. Corticosteroids are used as a pretreatment for infusion-related reactions or allergic reactions (e.g., medication before CT scans).

  (12) Pregnant or lactating women (13) Patients with currently uncontrolled comorbidities, such as decompensated cirrhosis, nephrotic syndrome, uncontrolled hyperglycemia, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, severe bleeding tendency, or coagulation disorders.

  (14) Patients with known allergies to any component of the study drug (oxaliplatin, capecitabine, QL1706); a history of severe allergic reactions to other monoclonal or bispecific antibodies; or known allergies to multiple substances or severe allergic diseases.

  (15) Patients who have received a live vaccine within 30 days prior to randomization or who plan to receive a live vaccine during the study period.

  (16) Patients with cognitive impairment or severe comorbid mental disorders, or those deemed by the investigator to have poor chemotherapy adherence; or other cases deemed unsuitable for participation in clinical trials by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | 1 year
  Complete response: Pathological complete response and clinical complete response

SECONDARY OUTCOMES:
R0 Resection Rate | 1 year
  The proportion of surgical patients who achieve an R0 resection. R0 resection: All gross disease has been removed, and microscopic examination reveals all surgical margins free of tumor.
Organ Preservation Rate (OPR) | 1 year
  The 1-year organ preservation rate is the percentage of patients attaining a complete clinical response (cCR) or near-complete clinical response (near-cCR) following neoadjuvant therapy, who then proceeded with non-surgical management or local excision, was monitored under a Watch & Wait strategy or for 1 year post-local resection without undergoing radical surgery.
Disease-free survival (DFS) | 3 years
  DFS is defined as the time from randomization to the earliest occurrence of any of the following events:
  Tumor progression by imaging according to RECIST 1.1, Tumor recurrence (local or distant), confirmed by imaging or biopsy, for patients with no residual tumor after surgery, Death from any cause. Note: A second primary malignancy is not considered an DFS event.
Overall survival (OS) | 3 years
  The time interval between the date of randomization to the date of death. If the patient has been alive, the time until the last follow-up is taken as the overall survival period.
Incidence of adverse events | During neoadjuvant chemoradiotherapy combined with immunotherapy, an average of 6 months
  Assessed by Common Terminology Criteria for Adverse Events version 4.0. The overall adverse event rates and the immune-related adverse event rates will be compared between treatment arms using Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No